CLINICAL TRIAL: NCT04418245
Title: Identification of Thoracic CT Scan Biomarkers by Deep Learning for Evaluating the Prognosis of Patients With COVID-19 Disease
Brief Title: CT Biomarkers Identification by Artificial Intelligence for COVID-19 Prognosis
Acronym: COVID 19-IA
Status: Withdrawn | Type: Observational
Why Stopped: Difficulties in setting up the study
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2020/COVID 19-IA/JF-01
Record Dates: First submitted 2020-06-04; First posted 2020-06-05 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Covid-19
Keywords: low dose CT scan; biomarkers; artificial intelligence
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients positive for SARS-CoV-2
  Interventions: Diagnostic Test: Imaging by thoracic scanner

INTERVENTIONS:
Diagnostic Test: Imaging by thoracic scanner — Low-dose computed tomography

SUMMARY:
The study hypothesis is that low-dose computed tomography (LDCT) coupled with artificial intelligence by deep learning would generate imaging biomarkers linked to the patient's short- and medium-term prognosis.

The purpose of this study is to rapidly make available an early decision-making tool (from the first hospital consultation of the patient with symptoms related to SARS-CoV-2) based on the integration of several biomarkers (clinical, biological, imaging by thoracic scanner) allowing both personalized medicine and better anticipation of the patient's evolution in terms of care organization.

ELIGIBILITY:
Inclusion Criteria:

* Patients positive for SARS-CoV-2 according to RT-PCR test between 1st March and 31st May 2020
* Patients undergoing low dose CT scan to establish Covid-19 lung damage
* Available for at least 8 days follow-up

Exclusion Criteria:

• Patients opposing the retrospective use of their data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized for Covid-19 confirmed by RT-PCR and undergoing CT scan
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Vital status | Day 8
  Dead/alive
Patient requiring more than 3 liters of oxygen to maintain a saturation >95% (intensive care unit or resuscitation department) | Day 8
  Yes/no
Percentage of lung affected on CT | Day 0
  % ground glass and condensation calculated by deep learning
Percentage of lung affected by ground glass opacity on scan | Day 0
  % calculated by deep learning
Percentage of lung affected by condensation on scan | Day 0
  % calculated by deep learning

SECONDARY OUTCOMES:
Vital status | Day 16
  Dead/alive
Vital status | Day 30
  Dead/alive
Length of hospitalization | Maximum 30 days
  Days
rehospitalization | Day 30
  Yes/no
Duration of intubation | Day 30
  Days
Percentage of lung affected on CT | Day 16
  % ground glass and condensation calculated by deep learning
Percentage of lung affected by ground glass opacity on scan | Day 16
  % calculated by deep learning
Percentage of lung affected by condensation on scan | Day 16
  % calculated by deep learning
Software operating time | End of study (August 2020)
  Speed of image loading and image processing depending of brand of scanner
C-reactive protein levels | Admission Day 0
  mg/L
lactate dehydrogenase | Admission Day 0
  U/L
lymphocytemia | Admission Day 0
  g/L
D Dimers level | Admission Day 0
  µg/L
Time until onset of symptoms | Admission Day 0
  Days
Time between RT-PCR positive results and first scan | Admission Day 0
  Hours
Age | Admission Day 0
  Years
BMI> 30 | Admission Day 0
  Yes/no:
Medical history of cardiovascular disease | Admission Day 0
  Yes/no: hypertension, coronary artery disease, congestive heart failure, cardiac arrhythmia
Diabetes | Admission Day 0
  Yes/no
Medical history of respiratory disease | Admission Day 0
  Yes/no: Chronic obstructive pulmonary disease, chronic respiratory failure
Medical history of immunosuppressed condition | Admission Day 0
  Yes/no: steroid use, pre-existing immunological condition, current chemotherapy for cancer
Current or previous history of smoking | Admission Day 0
  Yes/no:
Calculate a prognostic score from clinical, biological and CT parameters | Day 8
  Deep learning algorithm
Calculate a prognostic score from clinical and biological parameters only | Day 8
  Deep learning algorithm
Compare receiver operating curves of prognostic scores with and without CT parameters | Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Julien Frandon, Principal Investigator — CHU Nimes
Locations (6):
- France (5):
  - CHU la Timone, Marseille
  - CHU Montpellier, Montpellier
  - CHU de Nimes, Nîmes
  - CHU Poitiers, Poitiers
  - CHU Strasbourg, Strasbourg
- CHU Martinique, Fort-de-France, Martinique